CLINICAL TRIAL: NCT02946840
Title: The Use of a New Core Needle in the Endoscopic Ultrasound Assisted Tissue Sampling for Pancreatic Solid Masses
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Maggiore Bellaria Hospital, Bologna (Other); Catholic University of the Sacred Heart (Other); The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); Azienda Unità Sanitaria Locale di Imola (Other)
Responsible Party: Sponsor
Other Study IDs: Studio 1587
Record Dates: First submitted 2016-08-03; First posted 2016-10-27 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Pancreatic Masses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Solid pancreatic masses: Consecutive patients with solid pancreatic masses, submitted to FNA with 25 G Beacon needle (Medtronic, Newton, MA, USA)
  Interventions: Device: FNA with 25 G Beacon needle

INTERVENTIONS:
Device: FNA with 25 G Beacon needle

SUMMARY:
Endoscopic ultrasound-guided fine-needle aspiration biopsy (EUS-FNA) is a reliable, safe, and effective technique for obtaining samples from pancreatic masses. A new core biopsy needle has been developed by Beacon bnx® (Medtronic, Newton, MA) that allows the possibility to achieve a core for histology evaluation and the interchangibility of needle size using the same needle shelter and different needle sizes.

DETAILED DESCRIPTION:
At every pass, the material will be fixed in formalin. Three passes will be done. Details of the aspirated material will be described at macroscopic evaluation by the endoscopist and then by the pathologist at macroscopic and microscopic evaluation, in order to find an interobserved agreement on the definition of the core.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 and less than 90, both genders..
* Presence of a pancreatic solid lesion. In the presence of a cystic component, the solid part of the lesion should be more 75% of the total.
* Absence of an uncorrectable coagulopathy as defined by abnormal prothrombin time (PT) or partial thromboplastin time (PTT) that does not normalize after administration of fresh frozen plasma or coagulation factors.
* Informed consent is obtained.

Exclusion Criteria:

* Previous biopsy of the lesion with diagnosis of malignancy
* Presence of an uncorrectable coagulopathy as defined by abnormal prothrombin time (PT) or partial thromboplastin time (PTT) that does not normalize after administration of fresh frozen plasma.
* Pregnancy or breast-feeding.
* Patients unable to understand and/or read the consent form.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients referred for EUS examination and FNA of solid pancreatic masses, will undergo EUS-FNA with the 25G Shark core needle.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-08; Primary Completion 2017-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Core acquisition | 24 h
  The presence of a core adequate for histological evaluation for final diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, MD, Study Director — Humanitas University; Silvia Carrara, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan; Alberto Larghi, MD, Study Director — Università Cattolica
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Leo M, Crino SF, Bernardoni L, Rahal D, Auriemma F, Correale L, Donato G, Massidda M, Anderloni A, Manfrin E, Armellini E, Poliani L, Fugazza A, Semeraro R, Occhipinti P, Repici A, Carrara S. EUS-guided core biopsies of pancreatic solid masses using a new fork-tip needle: A multicenter prospective study. Dig Liver Dis. 2019 Sep;51(9):1275-1280. doi: 10.1016/j.dld.2019.03.025. Epub 2019 Apr 20. PMID 31010744